CLINICAL TRIAL: NCT01384097
Title: An Algorithm for Intra-operative Goal-directed Haemodynamic Management in Non-cardiac Surgery - a Feasibility Study
Brief Title: An Algorithm for Intra-operative Goal-directed Haemodynamic Management in Non-cardiac Surgery
Acronym: ERAS_feasi
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Department of Anesthesiology and Intensive Care Medicine CVK/CCM, Charite University, Berlin, Charite University, Berlin, Germany
Other Study IDs: ERAS_feasibility
Record Dates: First submitted 2011-06-27; First posted 2011-06-28 (Estimated); Last update posted 2011-09-08 (Estimated); Status verified 2011-09

CONDITIONS: Fracture of Surgical Neck of Humerus; Colonic Tumor; Stage IIIB Ovarian Carcinoma; Neoplasm of Head of Pancreas
Keywords: haemodynamic; goal-directed therapy; surgery; anaesthesia
MeSH Terms: conditions — Colonic Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Conventional care: patients treated by conventional haemodynamic care intraoperatively
- Haemodynamic algorithm: patients treated within a goal-directed haemodynamic algorithm intraoperatively

SUMMARY:
A systematic literature search a goal-directed haemodynamic algorithm was created. The hypothesis of this study was that the goal-directed haemodynamic algorithm is feasible and can improve clinical outcome.

DETAILED DESCRIPTION:
After a systematic literature search a goal-directed haemodynamic algorithm was created. The algorithm was adapted to international standards and consensus was reached through a modified Delphi method at international meetings. The feasibility of using the algorithm for intraoperative haemodynamic management was tested and the resultant clinical data analyzed retrospectively for several types of surgery with the hypothesis that the goal-directed haemodynamic algorithm is feasible in the clinical setting and can improve clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a surgical repair of hip fractures, open right hemicolectomy and extended hemicolectomy, radical tumor debulking in primary ovarian cancer or a pylorus-preserving pancreatic head resection at the Charité - University Medicine Berlin, Campus Virchow Clinic
* 18 years and older

Exclusion Criteria:

* emergency procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing a surgical repair of hip fractures, open right hemicolectomy and extended hemicolectomy, radical tumor debulking in primary ovarian cancer or a pylorus-preserving pancreatic head resection.
Sampling Method: Probability Sample
Enrollment: 774 (Actual)
Dates: Start 2007-09; Primary Completion 2011-02 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
hospital length of stay | a period of 60 days
  The perioperative hospital length of stay is assessed.

SECONDARY OUTCOMES:
need for ventilator therapy | a period of 60 days
  The perioperative need for ventilator therapy is assessed.
monetary reimbursement for prolonged hospital stay | a period of 60 days
  The monetary reimbursement for prolonged hospital stay is assessed to evaluate the impact on financial consequences.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD Prof., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité - University Medicine Berlin, Berlin, State of Berlin, Germany

REFERENCES:
- See also: The homepage of the Department of Anesthesiology and Intensive Care Medicine at the Charité - University Medicine Berlin — http://anaesthesieintensivmedizin.charite.de/